CLINICAL TRIAL: NCT05210413
Title: Spartalizumab and Low-dose PAzopanib in Refractory or Relapsed Solid TumOrs of Pediatric and Adults
Acronym: SPARTO
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: National Cancer Institute, France (Other Government); Fondation ARC (Other); Novartis (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2020/31
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Refractory or Recurrent Solid Tumor
Keywords: refractory or recurrent solid tumor; immunotherapy; modulators of angiogenesis
MeSH Terms: interventions — spartalizumab; pazopanib

STUDY DESIGN:
Intervention Model Description: Pediatric cohort:
  Multicentre, open-label, non-randomized, phase I clinical study, with dose-finding and expansion phases.
  Adult cohort:
  Multicenter phase II single-arm open-label clinical trial, with a pre-screening phase to identify patients with mature tertiary lymphoid structure (TLS).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pediatric cohort (Experimental): Multicentre, open-label, non-randomized, phase I clinical study, with dose-finding and expansion phases.
  Interventions: Drug: Spartalizumab in Pediatric cohort; Drug: Low-dose Pazopanib in Pediatric Cohort
- Adult cohort (Experimental): Multicenter phase II single-arm open-label clinical trial, with a pre-screening phase to identify patients with mature tertiary lymphoid structure (TLS).
  Interventions: Drug: Spartalizumab in Adult cohort; Drug: Low-dose Pazopanib in Adult Cohort

INTERVENTIONS:
Drug: Spartalizumab in Pediatric cohort — Infusion of spartalizumab at four dose escalation levels: 2, 3, 4 and 6 mg/kg in successive cohorts of 3 patients, depending on the number of patients with dose-limiting toxicity (DLT) to maximum tolerated dose (MTD).
  Arms: Pediatric cohort
Drug: Low-dose Pazopanib in Pediatric Cohort — Oral pazopanib treatment at a fixed dose of 225mg/m²/day
  Arms: Pediatric cohort
Drug: Spartalizumab in Adult cohort — Infusion of 400 mg of spartalizumab on Day1 of each cycle.
  Arms: Adult cohort
Drug: Low-dose Pazopanib in Adult Cohort — Oral pazopanib treatment with a fixed dose of 400 mg/day
  Arms: Adult cohort

SUMMARY:
Immunotherapies have revolutionized medical oncology following the remarkable and, in some cases, unprecedented outcomes observed in certain groups of patients with cancer. However results in adults and mainly in pediatric cancer are still disappointing.

Modulators of angiogenesis, such as VEGF, have a broad range of diverse effects on the immune system and the tumor micro-environment that are mainly immunosuppressive. In patients with early-stage disease, anti-VEGF therapy can lead to antitumor effects by modulating immune mechanisms - provided that therapy is maintained for an adequate length and tumors are sufficiently immunogenic. Nevertheless, blocking angiogenic molecules using a strategy based on a single therapeutic approach is likely insufficient to generate a complete or robust immune response against cancer, especially in patients with advanced-stage disease.

Based on the results of previous studies which evaluated the safety profile of spartalizumab, of pazopanib and the combination of antiangiogenic agents with checkpoint inhibitors, a study combining spartalizumab and low-dose pazopanib in refractory or relapsed solid tumors of pediatric and adults is proposed. This study will include 2 separate cohorts:

* the pediatric cohort will consist of a phase I study (dose-finding and expansion phases) combining pazopanib at a fixed dose of 225 mg/m2 and spartalizumab with four potential candidate doses (2, 3, 4 and 6 mg/kg).
* the adult cohort will consist of a phase II study combining pazopanib at a fixed dose of 400 mg and spartalizumab at the RP2D of 400 mg every 4 weeks.

DETAILED DESCRIPTION:
Immunotherapies have revolutionized medical oncology following the remarkable and, in some cases, unprecedented outcomes observed in certain groups of patients with cancer. However results in adults and mainly in pediatric cancer are still disappointing. One hypothesis is that the tumor micro-environment (TME) - characterized by hypoxia, a low pH, and a high interstitial fluid pressure - can reduce the effectiveness of virtually all types of anticancer therapies, including immunotherapy. In adults, combination with other therapeutic modalities, including anti-angiogenic agents, is one of the many strategies currently under investigation to improve the response rates and duration of immunotherapies.

Modulators of angiogenesis, such as VEGF, have a broad range of diverse effects on the immune system and the tumor micro-environment that are mainly immunosuppressive. In patients with early-stage disease, anti-VEGF therapy can lead to antitumor effects by modulating immune mechanisms - provided that therapy is maintained for an adequate length and tumors are sufficiently immunogenic. Nevertheless, blocking angiogenic molecules using a strategy based on a single therapeutic approach is likely insufficient to generate a complete or robust immune response against cancer, especially in patients with advanced-stage disease. Therefore, such anti-angiogenic agents will likely need to be used in combination with various immunotherapeutic strategies that boost adaptive immune responses, such as those described in the next sections. For these reasons, the investigators proposed to combine immunotherapy and low dose of pazopanib to enhance the efficacy of immunotherapy in some selected pediatric patients and adults.

PDR001 (also referred to as spartalizumab) is a humanized monoclonal antibody (mAb) directed against human programmed death-1 (PD-1) that blocks the interaction between PD-1 and its ligands (PD-L1 and PD-L2).

Pazopanib is a potent, selective, oral, ATP competitive multitargeted receptor tyrosine kinase inhibitor of vascular endothelial growth factor receptors (VEGFR) -1, -2, and -3, c-kit, and platelet-derived growth factor receptors. It is approved by the US Food and Drug Administration for the treatment of advanced renal cell carcinoma and soft tissue sarcoma (STS) in adults. Based on the results of previous studies which evaluated the safety profile of spartalizumab, of pazopanib and the combination of antiangiogenic agents with checkpoint inhibitors, a study combining spartalizumab and low-dose pazopanib in refractory or relapsed solid tumors of pediatric and adults is proposed. This study will include 2 separate cohorts:

* the pediatric cohort will consist of a phase I study (dose-finding and expansion phases) combining pazopanib at a fixed dose of 225 mg/m2 and spartalizumab with four potential candidate doses (2, 3, 4 and 6 mg/kg).
* the adult cohort will consist of a phase II study combining pazopanib at a fixed dose of 400 mg and spartalizumab at the RP2D of 400 mg every 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. For pediatric patients (Cohort 1):

   1. Patients should be without standard established therapeutic alternatives at the time of enrollment suffering from the following conditions :

      * refractory or recurrent solid tumor, proven histologically,
      * any tumor with high mutational load (> 10 somatic mutations/ Mo) or a high MSI status,
      * tumor, whatever the histology, with proven PDL1 expression (≥1%) or presence of mature tertiary lymphoid structure (TLS).
   2. Age ≥5 and <18 years at inclusion, patients 18 years and older may be included after discussion with the Sponsor if they have a pediatric recurrent/refacractory malignancy.
   3. Performance status: Karnofsky performance status (for patients >16 years of age) or Lansky Play score (for patients ≤16 years of age) ≥70%. Patients who are unable to walk because of paralysis or stable neurological disability, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
   4. Able to swallow tablets.
   5. Evaluable or measurable disease as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1…).
   6. Life expectancy ≥ 3 months.
   7. Adequate organ function:

      * Hematologic criteria :peripheral absolute neutrophil count (ANC) ≥1000/μL (unsupported), platelet count ≥100,000/μL (unsupported), hemoglobin ≥8.0 g/dL (transfusion is allowed)
      * Cardiac function: shortening fraction (SF) >29% (>35% for children <3 years) and left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography (mandatory only for patients who have received cardiotoxic therapy), absence of QTc prolongation (QTc >450 msec on baseline ECG, using the Fridericia correction [QTcF formula]) or other clinically significant ventricular or atrial arrhythmia.
      * Renal and hepatic function: serum creatinine ≤1.5 x upper limit of normal (ULN) for age, total bilirubin ≤1.5 x ULN, alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x ULN; aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT ≤ 2.5 x ULN except in patients with documented tumor involvement of the liver who must have AST/SGOT and ALT/SGPT ≤ 5 x ULN.
   8. Able to comply with scheduled follow-up and with management of toxicity.
   9. Females of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to initiation of treatment. Sexually active women of childbearing potential must agree to use a highly effective contraception during the study and for at least 6 months after the last study treatment administration. Sexually active male patients must agree to use condoms during the study and for at least 6 months after the last study treatment administration.
   10. Written informed consent from parents/legal representative and age-appropriate assent before any study-specific screening procedures are conducted according to local, regional or national guidelines.
   11. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.
2. For adults patients:

   * Pre-screening phase:

     1. adults (≥ 18 years old) with refractory or recurrent solid tumor (include rhabdomyosarcoma, Ewing's sarcoma, osteosarcoma and other) and/or tumor with High mutation rate (>10 somatic mutations/Mb) and/or suffering of Mismatch repair-deficient syndrome.
     2. Adult patients with an ECOG score of 0/1. Patients who are unable to walk because of paralysis or stable neurological disability, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
     3. Evaluable or measurable disease as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1…).
     4. Written informed consent from patient before any study-specific screening procedures are conducted according to local, regional or national guidelines.
   * Screening phase (Cohort 2):

     1. adults without standard established therapeutic alternatives at the time of enrollment suffering from refractory or recurrent advanced solid tumor characterized by the presence of mature TLS
     2. Age ≥ 18 years at inclusion
     3. Adult patients with an ECOG score of 0/1. Patients who are unable to walk because of paralysis or stable neurological disability, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.
     4. Evaluable or measurable disease as defined by standard imaging criteria for the patient's tumor type (RECIST v1.1…).
     5. Life expectancy ≥ 3 months
     6. Adequate organ function:
   * Hematologic criteria :peripheral absolute neutrophil count (ANC) ≥1000/μL (unsupported), platelet count ≥100,000/μL (unsupported), hemoglobin ≥8.0 g/dL (transfusion is allowed)
   * Cardiac function: shortening fraction (SF) >29% and left ventricular ejection fraction (LVEF) ≥50% at baseline, as determined by echocardiography (mandatory only for patients who have received cardiotoxic therapy), absence of QTc prolongation (QTc >450 msec on baseline ECG, using the Fridericia correction [QTcF formula]) or other clinically significant ventricular or atrial arrhythmia.
   * Renal and hepatic function: serum creatinine ≤1.5 x upper limit of normal (ULN) for age, total bilirubin ≤1.5 x ULN, alanine aminotransferase (ALT)/serum glutamic pyruvic transaminase (SGPT) ≤ 2.5 x ULN; aspartate aminotransferase (AST)/serum glutamic oxaloacetic transaminase/SGOT ≤ 2.5 x ULN except in patients with documented tumor involvement of the liver who must have AST/SGOT and ALT/SGPT ≤5 x ULN.

     g. Able to comply with scheduled follow-up and with management of toxicity. h. Females of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 72 hours prior to initiation of treatment. Sexually active women of childbearing potential must agree to use a highly effective contraception during the study and for at least 6 months after the last study treatment administration. Sexually active male patients must agree to use condoms during the study and for at least 6 months after the last study treatment administration.

     i. Written informed consent from patient before any study-specific screening procedures are conducted according to local, regional or national guidelines.

     j. Patient affiliated to a social security regimen or beneficiary of the same according to local requirements.

Exclusion Criteria:

For pediatric and adult patients (Cohorts 1 and 2):

1. Patients treated with anti-PD1 immunotherapy within 6 months prior to starting study treatment; patients treated with anti-PD1 for more than 6 months remain eligible for inclusion, provided that this treatment has brought the patient clinical benefit (objective response or stable disease > 4 months).
2. Impairment of gastrointestinal (GI) function or GI disease that may significantly alter drug absorption of oral drugs (e.g. ulcerative diseases, uncontrolled nausea, vomiting, diarrhea or malabsorption syndrome).
3. Clinically significant, uncontrolled heart disease (including history of any cardiac arrhythmia, e.g. ventricular, supraventricular, nodal arrhythmias, or conduction abnormality), unstable ischemia, congestive heart failure within 12 months of screening).
4. Uncontrolled hypertension
5. Active viral hepatitis or known human immunodeficiency virus (HIV) infection or any other uncontrolled infection.
6. Presence of any ≥ CTCAE grade 2 treatment-related toxicity with the exception of alopecia, ototoxicity or peripheral neuropathy.
7. Systemic anticancer therapy within 21 days of the first study dose or 5 times its half-life, whichever is less.
8. Previous myeloablative therapy with autologous hematopoietic stem cell rescue within 8 weeks of the first study drug dose
9. Allogeneic stem cell transplant within 3 months prior to the first study drug dose. Patients receiving any agent to treat or prevent graft-versus host disease (GVHD) post bone marrow transplant are not eligible for this trial.
10. Radiotherapy (non-palliative) within 21 days prior to the first dose of drug (or within 6 weeks for therapeutic doses of MIBG)
11. Major surgery within 21 days of the first dose. Gastrostomy, ventriculo-peritoneal shunt, endoscopic ventriculostomy, tumor biopsy and insertion of central venous access devices are not considered major surgery, but for these procedures, a 48-hour interval must be maintained before the first dose of the investigational drug is administered.
12. Currently taking medications with a known risk of prolonging the QT interval or inducing Torsades de Pointes
13. High dose chemotherapy followed by peripheral stem cell transplantation within less than 6 months.
14. Diagnosis of immunodeficiency or receiving systemic steroid therapy or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment. The use of physiologic doses of corticosteroids (up to 0.25 mg/kg daily prednisone equivalent) may be approved after consultation with the Sponsor.
15. Diagnosis of prior or active autoimmune disease.
16. Evidence of interstitial lung disease.
17. Unable to taper steroids due to ongoing mass effect; a maximum dexamethasone dose of 0.05 mg/kg/day is allowed, but preferably have been discontinued.
18. Known hypersensitivity to any study drug or component of the formulation.
19. Persons referred to in Articles L. 1121-5, L. 1121-6, L. 1121-8 and L. 11221-1-2 of the Public Health Code (pregnant women, parturient and nursing mothers; persons deprived of their liberty by a judicial or administrative decision, persons hospitalized without consent and persons admitted to a health or social establishment for purposes other than that of research; adults subject to a legal protection measure or incapacitated express consent; people in emergency situations who cannot give prior consent)
20. Vaccinated with live, attenuated vaccines within 4 weeks of the first dose of study drug.

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2025-08-26 (Actual); Study Completion 2027-11-17 (Estimated)

PRIMARY OUTCOMES:
The maximum tolerated dose (MTD) in the pediatric cohort | 2 months after inclusion ( treatment initiation)
  The maximum tolerated dose (MTD) in the pediatric cohort will be defined as the dose closest to the target toxicity level of 25% of DLTs (Dose Limiting Toxicity) up to cycle 2 (8 weeks of treatment).
  All patients will be evaluable for toxicity from the time of their first dose of study drug. All patients will be evaluable for DLT if they receive >75% of the planned dose after 2 cycles or if they have treatment-related toxicity at any time during the two cycles.
6-month disease control rate in the adult cohort | 6 months after inclusion ( treatment initiation)
  The 6-month disease control rate is defined as the proportion of participants in complete response (CR), partial response (PR) or stable disease (SD) 6 months after treatment initiation.
  All evaluable patients will be included in the response rate calculation. The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.

SECONDARY OUTCOMES:
Dose-limiting toxicity (DLT) in the pediatric cohort | 2 months after inclusion ( treatment initiation)
  A dose-limiting toxicity (DLT) is defined as a drug-related AE occurring in the first 8 weeks of study treatment.
  DLT will be defined as follows:
  * nausea, vomiting, alopecia, fever ≥ grade 3 lasting more than 72 hours
  * fatigue ≥ grade 3 lasting more than one week
  * other non-hematological toxicity ≥ grade 3
  * laboratory abnormality ≥ grade 3 lasting > 10 days (except for hyperglycaemia and changes in serum electrolytes/enzymes without clinical impact)
  * laboratory abnormality ≥ grade 4 (except for hyperglycaemia and changes in serum electrolytes/enzymes without clinical impact)
  * febrile neutropenia (ANC<1000/mm3 with a single temperature of >38.3 degrees C (101 degrees F) or a sustained temperature of >= 38degrees C (100.4 degrees F) for more than one hour)
  * grade 4 neutropenia lasting ≥ 10 days
  * grade 4 thrombocytopenia or grade 3 with bleeding requiring a platelet transfusion.
  * amylase or lipase elevation grade 3 with symptom or sign on imagery of pancreatitis
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] in pediatric and adult cohorts | 1 month after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 2 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 3 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 4 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 5 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 6 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 7 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 8 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 9 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 10 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 11 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]in pediatric and adult cohorts | 12 months after inclusion ( treatment initiation)
  Incidence of adverse events and serious adverse events, defined according to the NCI CTCAE v5.
Overall Response Rate in pediatric and adult cohorts | 12 months after inclusion ( treatment initiation)
  The best overall response is the best response (CR or PR) recorded from the start of the treatment until patients get off-study or the cut-off date, whichever comes first.
Progression-free survival in pediatric and adult cohorts | 12 months after inclusion ( treatment initiation)
  duration from start of the treatment to disease progression (clinically or radiologically) or death (regardless of cause of death), whichever comes first. Patients alive and free of progression at the cut-off date will be censored at the last assessment date.
Overall survival in pediatric and adult cohorts | 12 months after inclusion ( treatment initiation)
  duration from start of the treatment to death (regardless of cause of death). Patients alive at the cut-off date will be censored at the last assessment date
Response duration in pediatric and adult cohorts | 12 months after inclusion ( treatment initiation)
  Response duration will be measured from the time measurement criteria for CR/PR are first met until the first date that recurrent or progressive disease is objectively documented or death, whichever occurs earlier. Duration of response for patients free of progression at the cut-off date will be censored at the last imaging response-scan date.
Response rate in pediatric and adult cohorts | 2 months after inclusion ( treatment initiation)
  The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.
Response rate in pediatric and adult cohorts | 4 months after inclusion ( treatment initiation)
  The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.
Response rate in pediatric and adult cohorts | 8 months after inclusion ( treatment initiation)
  The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.
Response rate in pediatric and adult cohorts | 10 months after inclusion ( treatment initiation)
  The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.
Response rate in pediatric and adult cohorts | 12 months after inclusion ( treatment initiation)
  The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.
Response rate in pediatric cohort | 6 months after inclusion ( treatment initiation)
  The subjects that will be assigned a response category are all patients who have received at least one treatment dose and have had their disease reevaluated. Objective tumor response will be measured according to RECIST 1.1 (Eisenhauer 2009) for solid tumor.

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane DUCASSOU, MD, PhD, Principal Investigator — University Hospital, Bordeaux
Locations (13):
- France (13):
  - CHU d'Angers - Unité d'Hématologie et d'Oncologie pédiatrique, Angers
  - CHU de Bordeaux - Unité d'Hématologie et d'Oncologie pédiatrique, Bordeaux
  - Institut Bergonié - Oncologie Médicale, Bordeaux
  - Centre Oscar Lambret - Oncologie pédiatrie, Lille
  - Oscar Lambret Center, Lille
  - Centre Léon Bérard - Oncologie Médicale, Lyon
  - Institut d'Hématologie et d'Oncologie Pédiatrique (IHOP) - Oncologie pédiatrique, Lyon
  - APHM Hôpital des Enfants La Timone - Hématologie Oncologie Pédiatrique, Marseille
  - Nantes University Hospital, Nantes
  - Institut Curie - Centre D'Oncologie SIREDO, Paris
  - Curie Institute, Paris
  - Strasbourg University Hospital, Strasbourg
  - Gustave Roussy - Oncologie pédiatrique, Villejuif

IPD SHARING:
Plan to Share IPD: No